CLINICAL TRIAL: NCT02761798
Title: The Automated Mobile Interactive Audiometer - Feasibility and Reliability in a Clinical Setting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Matt Bromwich (Other)
Collaborators: Clearwater Clinical (Unknown); Children's Hospital of Eastern Ontario (Other)
Responsible Party: Sponsor-Investigator, Matt Bromwich, Otolaryngologist, Head and Neck Surgeon, Ottawa Hospital Research Institute
Organization: Ottawa Hospital Research Institute (Other)
Other Study IDs: 20150561-01H
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Automated Mobile Interactive Audiometer, Test Retest: Each participant will act as his/her own control. The iPad audiogram will be compared to the audiogram in sound booth or to a second iPad audiogram.
  Interventions: Device: Automated Mobile Interactive Audiometer
- Automated Mobile Interactive Audiometer, Validation.: iPad testing will be compared to conventional audiometry in the sound booth.
  Interventions: Device: Automated Mobile Interactive Audiometer
- Automated Mobile Interactive Audiometer, Speech Recognition: Testing with NU-6 word lists will be conducted by the iPad and by an audiologist in the sound booth.
  Interventions: Device: Automated Mobile Interactive Audiometer
- Automated Mobile Interactive Audiometer, Cochlear Implant: Participants with cochlear implants will be tested using iPad against conventional audiometry (warble tone) in the sound booth.
  Interventions: Device: Automated Mobile Interactive Audiometer

INTERVENTIONS:
Device: Automated Mobile Interactive Audiometer — iPad game

SUMMARY:
This observational study aims to validate the use of a tablet based audiometer to provide an accurate, efficient, and cost-effective means for diagnosis of hearing conditions in controlled and uncontrolled environments in adult and elderly populations.

DETAILED DESCRIPTION:
In the 2011 report on Disability, the World Health Organization rated hearing loss as the most prevalent disability in the world. More than 30% of adults have disabling hearing loss complicating the management of their comorbid diseases. Isolation, mental illness and lack of family support are just some of the negative impacts of this invisible disability. In the next 25 years the number of hearing impaired individuals over the age of 65 in Canada will double, while at the same time there is a projected 50% shortfall in audiological service providers. The resultant service deficit is compounded by the lack of equipment and familiarity with hearing healthcare at the primary care level, causing increased inefficiency, unnecessary referrals, and unmet needs.

In Canada, there is a critical need to improve the number of health professionals with the requisite skills to meet the needs of the aging population. This project is aimed at developing a novel approach to address the increasing need for hearing healthcare in the adults while managing the strain on the healthcare system.

Healthcare workers (such as general practitioners, registered nurses and allied heath workers) can play an important role in supporting and motivating adults to seek help and aid in the referral process. However, few healthcare workers receive formal training in the identification, diagnosis, treatment options, referral process, and special needs of older adults with hearing loss. This lack of training, resources and equipment is a significant gap in the care provided to the elderly and impacts all other aspects of elder care.

Undiagnosed/untreated hearing loss can lead to physiological changes associated with auditory deprivation, as well as psychosocial changes of social isolation and depression. It can result in emotional, physical, cognitive, and behavioral consequences including impaired activities of daily living, decline in independence and reduced quality of life. In spite of the prevalence and impact of hearing loss and the benefits of rehabilitation in reducing the psychological, social, and emotional consequences of hearing loss, referral by physicians for assessment and rehabilitation is low and the majority of adults who could benefit from the use of hearing aids do not use this technology. Early identification can help to reduce these deleterious effects, and lead to easier adjustment to hearing aid use.

In spite of the numerous recent technological advances in field of hearing amplification devices, current technologies may not be effective for older adults who have central auditory processing and cognitive processing difficulties. Additionally, untreated hearing loss lowers performance on aurally administered diagnostic tests used to quantify the severity of dementia and can significantly confound the clinical picture in this population. Furthermore, the use of amplification is associated with reduction in problem behavior in persons with a primary diagnosis of Alzheimer's disease and a reduction in hearing handicap for persons with Alzheimer's disease and their significant others.

This study aims to validate the use of a tablet based audiometer to provide an accurate, efficient, and cost-effective means for diagnosis of hearing conditions in controlled and uncontrolled environments in adult and elderly populations.

Observations between the soundbooth and iPad audiograms will include the following frequencies 250, 500, 1000, 2000, 4000, 6000 and 8000 Hz. Each iPad audiogram consists of an interactive game that takes approximately 10-20 minutes to complete. The conventional audiogram will take place before the iPad audiogram. We expect our study to add a maximum of 20-30 minutes to each enrolled patient's visit. The iPad audiogram observations will not be used by the patient's physician for diagnostic and treatment purposes.

ELIGIBILITY:
Inclusion Criteria:

* For Group I and II all adults over the age of 18 years who attend an Audiology clinic for conventional Audiometry at the Civic campus will be eligible for this study.
* For Group III adults over the age of 18 years who attend ENT clinic but aren't undergoing conventional audiometric testing will be eligible.

Exclusion Criteria:

* Patients who self report being unable to play the iPad game.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (> or equal to18 years) attending the ENT/Audiology clinic at The Ottawa Hospital (CIVIC Campus) will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Validate the use of an iPad audiometer for hearing testing in adults aged 18 and older in Ottawa, Canada. | 8 months
  iPad audiogram will be compared to conventional audiogram (sound booth) and test/retest reliability of the iPad will be measured in Group 3.

CONTACTS AND LOCATIONS:
Overall Officials: David Schramm, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Civic and General Campuses, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bastianelli M, Mark AE, McAfee A, Schramm D, Lefrancois R, Bromwich M. Adult validation of a self-administered tablet audiometer. J Otolaryngol Head Neck Surg. 2019 Nov 7;48(1):59. doi: 10.1186/s40463-019-0385-0. PMID 31699157